CLINICAL TRIAL: NCT03493295
Title: Non-interventional, Real Life Study on Satisfaction With LNG-IUS in Spanish Young Women (18-30 Years Old) With Different Parity Status and Menstrual Bleeding Pattern
Acronym: BERTA
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 19704
Record Dates: First submitted 2018-04-04; First posted 2018-04-10 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Contraception

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Levonogestrel IntraUterine System (LNG-IUS): Women in childbearing age between 18 to 30 years old and who have freely chosen a LNG-IUS for contraception after being adequately counselled and informed of all contraceptive options by their physician at the routine clinical practice setting in Spain
  Interventions: Drug: Levonogestrel IntraUterine System (LNG-IUS)

INTERVENTIONS:
Drug: Levonogestrel IntraUterine System (LNG-IUS) — At the routine clinical practice. Jaydess, Mirena, Kyleena Or any other levonogestrel intrauterine system (LNG-IUS) commercialized in Spain at the start of the study, only for contraception indication.

SUMMARY:
The aim of this non-interventional study (NIS) is to assess, under real-life conditions, woman's satisfaction with Levonogestrel IntraUterine System (LNG-IUS) in a young (18-30 years old (y.o.)) Spanish population taking into account their parity status.

Furthermore, the study is aimed to evaluate the impact of: menstrual bleeding pattern and satisfaction with it at baseline, LNG-IUS chosen, previously used contraceptive method and reasons for change to/ choice of a LNG-IUS on overall satisfaction with LNG-IUS use.

ELIGIBILITY:
Inclusion Criteria:

* Women in childbearing age, between 18-30 years old.
* Women who have chosen a LNG-IUS as contraceptive method, after been adequately counselled by the physician about all contraceptive possible options.
* Women who have chosen a LNG-IUS mainly for contraceptive reasons, not due to heavy menstrual bleeding.
* Women with no desire to conceive for at least within the next 12 months.
* Women capable of reading and writing

Exclusion Criteria:

* Women whose main reason to use a LNG-IUS is not a contraceptive reason.
* Women with contraindication for LNG-IUS.
* Women with previous experience with a IUS.
* Women who have been diagnosed with heavy menstrual bleeding.
* Women with degenerative or other kind of diseases that could directly negatively impact their daily life.
* Women who have undergone a hysterectomy or irreversible contraceptive method.
* Women participating in a clinical trial.
* Women with a mental illness and unable to make decisions and follow instructions.
* Women with amenorrhea
* Women with clinical history of severe dysmenorrhea
* Women with concomitant medication that may lead changes in bleeding pattern (e.g. antiplatelets and/or anticoagulants)

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants will be women in childbearing age between ≥18 to 30 years, who have freely chosen a LNG-IUS for contraception after being adequately counselled and informed of all contraceptive options by their physician at a routine visit prior to the first study visit (enrolment) in a routine clinical practice setting. Then, women eligible for the enrolment will be visiting the physician in a IUS insertion visit in a gynaecological clinical setting.
Sampling Method: Non-Probability Sample
Enrollment: 587 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects rating 1 (very dissatisfied) to 5 (very satisfied) in the 5-point Likert scale overall satisfaction with LNG-IUS | At approximately 12 months(end of observation/final visit)
  Overall satisfaction with LNG-IUS at end of observation/final visit (i.e. after approximately 12 months or at premature discontinuation). 5 point Likert scale of overall satisfaction with LNG-IUS with end labelling "very dissatisfied" / "very satisfied"

SECONDARY OUTCOMES:
Percentage of women rating 1 (very dissatisfied) to 5 (very satisfied) in the 5-point Likert scale of overall satisfaction with the menstrual bleeding profile with LNG-IUS | At 4-12 weeks after insertion, At approximately 12 months(end of observation/final visit)
  Overall satisfaction rate with LNG-IUS at end of observation/final visit. 5 point Likert scale of overall satisfaction with the menstrual bleeding pattern with LNG-IUS with end labelling "very dissatisfied" / "very satisfied".
8 item user satisfaction questionnaire to assess the satisfaction with menstrual bleeding pattern with LNG-IUS | At approximately 12 months(end of observation/final visit)
  Overall satisfaction with the menstrual bleeding profile with LNG-IUS at end of observation/final visit.
Spearman's correlation between overall satisfaction with LNG-IUS and overall satisfaction with menstrual bleeding pattern | At approximately 12 months(end of observation/final visit)
Percentage of subjects rating 1 (very dissatisfied) to 5 (very satisfied) in the 5-point Likert scale overall satisfaction with LNG-IUS | At 4-12 weeks after insertion
  Overall satisfaction with LNG-IUS 4-12 weeks after insertion. 5 point Likert scale of overall satisfaction with LNG-IUS with end labelling "very dissatisfied" / "very satisfied"
Overall satisfaction with the menstrual bleeding profile 4-12 weeks after insertion. | At 4-12 weeks after insertion
Ease of LNG-IUS insertion will be measured by investigator on an ordinal scale of "easy", "slightly difficult", "very difficult" | At initial visit (Day 0_LNG-IUS insertion)
  Ease of LNG-IUS insertion assessed by the investigator.
Pain at LNG-IUS insertion will be assessed by the clinician asking to the user on a ordinal scale of "none", "mild", "moderate" or "severe" | At initial visit (Day 0_LNG-IUS insertion)
  Pain at LNG-IUS insertion assessed by the user.
Percentage of women that would recommend a LNG-IUS to peers | At approximately 12 months
  Response in recommendation to peers item at final visit.
Reasons for change to/ choice a LNG-IUS assessed by a multiple choice item | At initial visit (Day 0_LNG-IUS insertion)
Descriptive analysis of demographic data | At initial visit (Day 0_LNG-IUS insertion)
  Women's profile defined by their sociodemographic and gynaecological characteristics.
Reasons for withdrawal | Up to approximately 12 months
Percentage of withdrawal | Up to approximately 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Many locations, Multiple Locations, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- [Background] Perello Capo J, Lopez Gonzalez G, Rius-Tarruella J, Calaf Alsina J. Real-world satisfaction and menstrual bleeding pattern with available LNG-IUD among Spanish young women. Eur J Contracept Reprod Health Care. 2022 Dec;27(6):461-472. doi: 10.1080/13625187.2022.2112562. Epub 2022 Sep 23. PMID 36148980
- See also: Click here to find results for studies related to Bayer products. — http://clinicaltrials.bayer.com/